CLINICAL TRIAL: NCT01032941
Title: A Randomized Controlled Trial on the Beneficial Effects of Probiotics on Portal Hemodynamics in Decompensated Cirrhotic Patients
Brief Title: The Effect of Probiotics (VSL) on Portal Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Puneeta Tandon, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: VSL3PHTNUoA
Record Dates: First submitted 2009-12-03; First posted 2009-12-16 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Portal Hypertension
Keywords: Portal Hypertension; Portal Pressure Measurement; VSL3; Cirrhosis; End Stage Liver Disease; Probiotics
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; End Stage Liver Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in this group will be given placebo 2 packets BID for 8 weeks.
  Interventions: Drug: Probiotic
- VSL#3 (Experimental): Patients in this group will be given 2 packets of VSL#3 BID for 8 weeks.
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — Patients in this group will be given the probiotic VSL#3 2 packets BID for a total of 8 weeks.
  Other Names: VSL#3

SUMMARY:
The investigators will address the hypothesis that portal hypertension is mediated in part by bacterial or endotoxin translocation and the production of inflammatory mediators (tumor necrosis factor-α (TNFα), etc.). The investigators hypothesize that food supplementation with the probiotic product VSL#3 in patients with Child Pugh B/C cirrhosis will have a beneficial effect on in portal pressure (as measured by the HVPG) by reducing inflammatory mediators and improving systemic and splanchnic hemodynamics.

DETAILED DESCRIPTION:
We have recently completed an open-label uncontrolled trial of the probiotic VSL#3 in 8 patients with compensated cirrhosis and evidence of portal hypertension (VIP study) to determine whether this agent would have beneficial effects in portal pressure reduction (unpublished data Tandon, P. et al.). The open label design and the inclusion of compensated (Child Pugh A) cirrhotic patients in this initial study were chosen to confirm the safety and tolerance of VSL#3 and the safety of the portal pressure measurements at our center. No changes of physical status occured. There was a non-significant reduction in portal pressure from 19.7 to 18.1 mm Hg after 2 months of VSL#3 supplementation. Furthermore, there was a significant reduction in the serum aldosterone level (p=0.03). IL-8 levels were reduced in 4/6 patients analyzed to date. These results suggest that VSL#3 results in cytokine reduction and an improvement in the effective circulating volume even in these well-compensated cirrhotic patients. The comparison of the rest of the pro-inflammatory mediators and stool microflora is still being analyzed.

The data in our initial study is very promising. As our patients were compensated cirrhotics with normal intestinal permeability and only mild baseline perturbations in hepatic function parameters (INR, bilirubin, albumin) and neurohormonal markers (aldosterone, renin), it is not surprising that a reduction in portal pressure was not identified. Consistent with previous studies however, these local results confirm the safety and tolerance of both VSL#3 as well as portal pressure measurements in cirrhotic patients (20,24,25).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Cirrhosis
* Childs-Pugh Class B/C

Exclusion Criteria:

* Bacterial infection
* Grade 3-4 hepatic encephalopathy
* GI bleeding in the past 2 weeks
* Hepatocellular carcinoma beyond the Milan criteria
* Transjugular intrahepatic portosystemic shunt (TIPS), surgical shunt
* Portal vein thrombosis
* Antibiotics in the past 2 weeks
* Myocardial infarction, stroke or life-threatening arrhythmia within the last 6 months
* Active alcohol or illicit drug use
* Failure to consent to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction in portal pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, MD, FRCPC, MSc, Principal Investigator — University of Alberta; Vince Bain, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada